CLINICAL TRIAL: NCT05377463
Title: Optimizing a Bio-behavioral Intervention to Promote Viral Suppression Among HIV+ People Who Inject Drugs on the U.S.-Mexico Border
Brief Title: Optimizing a Bio-behavioral Intervention for Sustained Viral Suppression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Collaborators: University of California, San Francisco (Other); Centro de Integracion Juvenil (Unknown); El Centro Ambulatorio para la Prevención y Atención en SIDA e Infecciones de Transmisión Sexual (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1780619-1
Record Dates: First submitted 2022-04-11; First posted 2022-05-17 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: HIV Viremia
Keywords: HIV viral suppression
MeSH Terms: interventions — glycine N-choloyltransferase

STUDY DESIGN:
Intervention Model Description: The factorial experiment is guided by the Multiphase Optimization Strategy (MOST).
  The 2 intervention components are:
  Component 1. Peer recovery coaching to promote uptake and persistence of medication assisted treatment in the form of methadone.
  Component 2. Behavioral activation therapy to reduce depression.
  Participants will be randomly assigned to receive a total of 0 or up to 2 components. There are 4 conditions because there are 4 possible combinations of the 2 components (e.g., Condition 1 = Delivery of 1 whereas Condition 3 = Delivery of 1 and 2). All participants will receive a standard of care package which will consist of referral and patient navigation to HIV treatment services, linkage to a peer support group, and harm reduction education and materials.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blind to the experimental condition that the participant was assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1: Component 1 (Experimental): 1) Peer-Support for Medication-Assisted Treatment
  Interventions: Behavioral: Peer support to promote uptake and persistence of medication assisted treatment (MAT)
- Condition 2: Component 2 (Experimental): 2) Behavioral Activation Therapy
  Interventions: Behavioral: Behavioral Activation Treatment (BAT) to reduce depression
- Condition 3: Components 1 and 2 (Experimental): Participants assigned to a combination of:
  1. Peer-Support for Medication-Assisted Treatment
  2. Behavioral Activation Therap
  Interventions: Behavioral: Peer support to promote uptake and persistence of medication assisted treatment (MAT); Behavioral: Behavioral Activation Treatment (BAT) to reduce depression
- Condition 4: No Components (Experimental): Participants not assigned to any of the 2 components. They are placed on a wait list and will receive components after the primary data collection period.
  Interventions: Behavioral: No Intervention Components

INTERVENTIONS:
Behavioral: Peer support to promote uptake and persistence of medication assisted treatment (MAT) — Participants will be assigned to receive peer support to promote uptake of MAT and persistence. This component will consist of two informational sessions, a tailored recovery plan, and on-going support from a peer for the first 6 months.
  Arms: Condition 1: Component 1; Condition 3: Components 1 and 2
Behavioral: Behavioral Activation Treatment (BAT) to reduce depression — Participants will be assigned to receive BAT treatment for depression. This component will consist of 8 sessions where participants will identify short and long-term goals, values, and the activities unrelated to substance use that were previously enjoyed or are likely to increase a feeling of well-being. This intervention component focuses on making a plan to troubleshoot barriers to re-engage in these activities. Sessions are delivered weekly. The content includes psycho-education about what depression is, the intervention rationale, and the activities and monitoring of activities, building social contracts to engage networks, and discussion of potential barriers to following through with activities.
  Arms: Condition 2: Component 2; Condition 3: Components 1 and 2
Behavioral: No Intervention Components — Participants not assigned to components 1 and 2
  Arms: Condition 4: No Components

SUMMARY:
The study will test two behavioral intervention components to identify the combination of the two components that best supports people who inject drugs to achieve and sustain HIV viral load suppression.

The study design is a 2-to-the-2 factorial experiment. The 2 represents the level of each component: 0 (receive) or 1 (don't receive). The 2 represents the number of components being tested. The four components are: 1) receiving (or not receiving) peer support services for medication-assisted treatment (MAT) uptake and persistence and 2) behavioral activation therapy for depression (BAT). Therefore, in order to test which combination of components produce the best outcome, this factorial design randomizes people to 1 of 4 conditions. Each condition represents a possible combination of the 2 components above. All participants will receive patient navigation for care engagement.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of 4 experimental conditions. Each condition will represents every possible combination of 2 components (e.g., 1 only, 2 only, 1-2, none). Participants complete a survey assessment at baseline, complete their assigned intervention components, and then return to complete follow-up assessment surveys at 3-, 6-,9-, and 12-months. The primary outcome is sustained viral suppression defined as viral load test results of <400 copies per mL on all 6-,9-, and 12-month follow-up visits. Results of Aim 1 will yield estimates of the unique impact of each intervention component, as well as each combination of components, on sustained viral suppression. The research team and partners will make decisions about what constitutes the optimized intervention by judging the observed effect sizes and statistical significance against real-world constraints that go into the delivery of the interventions. The secondary aims are to test mediators to explain component 1-2 and its relationship to viral suppression. We will also test moderators of these relationship between each component and outcome of viral suppression.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* be able to provide informed consent
* be eligible to receive free HIV care services in Mexico
* be HIV positive
* have injected drugs in the last 30 days
* not be on methadone replacement therapy
* be willing to discuss MAT uptake with a peer
* sign a medical release form to have medical data abstracted
* agree to submit and describe locator information
* agree to return to follow-up visits
* able to communicate in Spanish
* screen positive for depression on the PHQ-2
* have no plans of moving outside the study area in the next 12-months
* meet one of the following:

  1. not currently in possession of ART or not taking ART but prescribed ART or
  2. sub-optimal ART adherence as at least one 4-day treatment interruption in the past 90 days or
  3. sub-optimal retention in HIV care - never engaged or disengaged from HIV care as 2 or more missed clinic appointments in the last 9 months or
  4. no viral load test done in the past six months or
  5. self-reports a detectable viral load within the past 6 months

Exclusion Criteria:

* has not injected drugs in the last 30 days or do not have a verifiable opioid use disorder
* is not HIV positive
* is receiving methadone
* is unwilling to discuss methadone uptake with a peer
* does not screen positive for depression
* is not able to provide informed consent
* does not speak Spanish
* has plans to move out of the city
* does not qualify to receive free HIV care services in Mexico
* has an appearance of psychological disturbance or severe cognitive impairment that could limit understanding of study procedures as determined by study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of Viral Suppression | Viral load below or above 400 copiers per mL at the 6-month follow-up assessment
  Viral suppression is defined as a laboratory test result showing HIV viral load as less than 400 copies per mL. To meet our definition of achieved viral suppression, viral load must be below 400 copiers per mL at 6-month follow-up.
Viral Suppression at 9-month follow-up | Viral load below or above 400 copiers per mL at the 9-month follow-up assessment
  Viral suppression is defined as a laboratory test result showing HIV viral load as less than 400 copies per mL. To meet our definition of viral suppression, viral load must be below 400 copiers per mL at 6-month follow-up.
Viral Suppression at 12-month follow-up | Viral load below or above 400 copiers per mL at the 12-month follow-up assessment
  Viral suppression is defined as a laboratory test result showing HIV viral load as less than 400 copies per mL. To meet our definition of viral suppression, viral load must be below 400 copiers per mL.

SECONDARY OUTCOMES:
Drug use | 3-,6-,9-, and 12-month follow-up assessments
  Will be measured through urine analysis and participants will self-report the frequency (yes vs no), quantity (how much typically consumed when using), and duration of use (how may days in the last 30 days did the participant use and how many times did the participant use yesterday) of various drugs in last 30 days.
Methadone uptake and persistence | 3-,6-,9-, and 12-month follow-up assessments
  Information about date of first dose, current dosage, and number of days on Methadone will be extracted from the medical record.
Drug use frequency and severity of withdrawal and cravings | 3-,6-,9-, and 12-month follow-up assessments
  Opioid Withdrawal Scale - This is a clinician administered scale that assesses the extent opiate withdrawal symptoms based on 11 symptoms (resting pulse rate, sweating, restlessness, pupil size, bone or joint aches, runny nose, GI upset, tremors, yawning, anxiety or irritability, gooseflesh skin.
Depressive Symptoms (Clinician-assisted rating) | 3-,6-,9-, and 12-month follow-up assessments
  The Montgomery-Asberg Depression Rating Scale will be used, which is a 10-item scale and is clinician-assisted. interview participants and clinicians will rate their level of depression. Symptoms assessed include: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts
Depressive Symptoms (Self-report) | 3-,6-,9-, and 12-month follow-up assessments
  The validated nine-item patient health questionnaire will be administered to participants to measure their level of depression. Participants will be asked to rate how many days of the last 2 weeks they have been bothered by having little interest or pleasure doing things, feeling down, feeling tired, having poor appetite, feeling bad about themselves, having trouble concentrating, moving or speaking slowly, and having thought of hurting themselves.
Behavioral activation for depression | 3-,6-,9-, and 12-month follow-up assessments
  The validated 25 item questionnaire will be administered to participants to assess changes in the behaviors in the past week that underlie their depression such as staying in bed too long, inability to do things that needed to be done, and being active and accomplishing goals.
Adherence to antiretroviral medication (ART) | 3-,6-,9-, and 12-month follow-up assessments
  Percent adherent to ART measure will be extracted from medical records
Non-adherence to antiretroviral medication (ART) | 3-,6-,9-, and 12-month follow-up assessments
  Non-adherence will be measured as 4-day treatment interruptions (yes vs no) extracted from medical records.
Information, motivation, and behavioral skills to adhere to ART | 3-,6-,9-, and 12-month follow-up assessments
  Participants will answer the validated 30-item scale to assess psychological precursors of adherence including information (e.g., knowledge of how current HIV medications should be taken); Motivation (e.g., support from close significant others to take HIV medication); Behavioral skills (e.g, how easy it is to get HIV medications refills on time)
Self-efficacy to adhere to ART | 3-,6-,9-, and 12-month follow-up assessments
  Participants will answer the validate 12-items scale assessing perceived self-efficacy to adhere to antiretroviral medication in the last 30 days. The scale asks about the level of confidence the participant has in keeping up with the treatment plan in spite of difficulties such as sided-effects and amid change in sleep and dietary habits and ability to integrate taking medications into the daily routine
Retention in HIV care | 3-,6-,9-, and 12-month follow-up assessments
  Retention will be assessed by extracting from the medical record: appointments missed and appointments kept. A ratio will be computed using these two measures. At least one appointment kept in each three-month period will be an index of appointment constancy.
Logistical barriers to HIV care | 3-,6-,9-, and 12-month follow-up assessments
  Participants will be asked to indicate whether they have experienced common barriers to HIV care (yes/no) including availability of transportation, being able to access care, clinic hours of operation.
Perceived engagement in HIV care | 3-,6-,9-, and 12-month follow-up assessments
  Participants will answer the 10-item validated scale assessing perceived engagement in HIV care including level of trust in provider, feeling respected and understood by provider, degree of comfort in asking questions and interacting with provider, participant's perceived role in his medical care,.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lechuga, Principal Investigator — The University of Texas at El Paso; John A Sauceda, Principal Investigator — The University of California San Francisco
Locations (1):
- Programa Compañeros, Ciudad Juárez, Chihuahua, Mexico

IPD SHARING:
Plan to Share IPD: Yes
We will share a final modified quantitative dataset with the corresponding code book to validate all findings. The dataset will be modified to remove any potential identifiable information (such as date of birth).
  Interested parties will be asked to sign an agreement with MPIs Lechuga and Sauceda that specifies that the use of the data is for research purposes only. Furthermore, in order to have the data shared, each party must have: a) adequate systems in place to secure, encrypt and protect the data file to prevent the disclosure of identities, and b) a plan for destruction or returning the data files after all analyses have been completed. Prior to the sharing of data, approval from the requester's Institutional Review Board is required.
Time Frame: The data will be made available as soon as possible but no later than within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier.
Access Criteria: Directions for requesting the dataset will be available at the official study website, which is to be developed. This information will be found in all publications and conference abstract presentations. An individual participant data statement noting steps to access the data is to be developed.

REFERENCES:
- [Derived] Sauceda JA, Lechuga J, Ramos ME, Puentes J, Ludwig-Barron N, Salazar J, Christopoulos KA, Johnson MO, Gomez D, Covarrubias R, Hernandez J, Montelongo D, Ortiz A, Rojas J, Ramos L, Avila I, Gwadz MV, Neilands TB. A factorial experiment grounded in the multiphase optimization strategy to promote viral suppression among people who inject drugs on the Texas-Mexico border: a study protocol. BMC Public Health. 2023 Feb 10;23(1):307. doi: 10.1186/s12889-023-15172-2. PMID 36765309

DOCUMENTS (1):
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05377463/ICF_000.pdf